CLINICAL TRIAL: NCT01104519
Title: A Randomized, Double-Blind, Placebo-Controlled, 2-Period Crossover Study to Evaluate the Effects of Multiple Oral Doses of 2000 mg of Niaspan on Endothelium-Dependent and Endothelium-Independent Vascular Reactivity in Subjects With Hypercholesterolemia
Brief Title: A Study of Niaspan on Endothelium-Dependent and Endothelium-Independent Vascular Reactivity (0000-093)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-093; 093; 2010_524
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Niaspan - Placebo
  Interventions: Drug: Niaspan; Drug: Comparator: Placebo
- 2 (Experimental): Placebo - Niaspan
  Interventions: Drug: Niaspan; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Niaspan — Oral doses of 2000 mg of Niaspan once daily for 7 days.
Drug: Comparator: Placebo — Oral doses of placebo once daily for 7 days.

SUMMARY:
A study to evaluate the inter- and intra subject variabilities of flow-mediated dilation (FMD) of brachial artery and nitroglycerin (GTN) induced dilation of brachial artery.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of reproductive potential test negative for pregnancy and agree to use appropriate methods of contraception throughout the study
* Subject is in good health (other than history of high cholesterol)
* Subject is a non-smoker

Exclusion Criteria:

* Subject has a history of stroke, seizures or major neurological disorder
* Subject has a history of cancer
* Subject is unable to refrain from or anticipates the use any prescription or non-prescription drugs
* Subjects consumes excessive amounts of alcohol or caffeine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
flow-mediated dilation (FMD) of brachial artery | predose, 4 hours post dose and 24 and hours post dose
Nitroglycerin (GTN) induced dilation of brachial artery | predose, 4 hours post dose and 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC